CLINICAL TRIAL: NCT07228377
Title: Digital Intervention for Symptom Management in Cancer and Opioid Sparing Using Virtual Reality (DISCOVR) - Feasibility, Acceptability, Usability Testing of a Novel Intervention
Brief Title: Digital Intervention for Symptom Management in Cancer and Opioid Sparing Using Virtual Reality (DISCOVR) Study
Acronym: DISCOVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00010075; 1R43CA302795-01A1 (NIH)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: cancer pain; chronic pain; opioid; virtual reality; technology
MeSH Terms: conditions — Neoplasms; Cancer Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality pain therapy (Experimental)
  Interventions: Behavioral: virtual reality pain therapy

INTERVENTIONS:
Behavioral: virtual reality pain therapy — DISCOVR virtual reality pain therapy

SUMMARY:
Patients living with cancer commonly have chronic pain due to the disease or to cancer treatments. Virtual reality, a new technology that immerses the user in pleasant, diverting, and exciting virtual environments, may lower chronic cancer pain to improve quality of life and complement need for pain medications like opioids. The investigators aim to learn from patients about the experience of cancer pain, develop a virtual reality prototype specific to cancer pain management, and test the feasibility and acceptability of this technology to improve the cancer pain experience.

DETAILED DESCRIPTION:
Patients living with cancer commonly experience chronic pain, defined as pain lasting at least three months. While cancer pain management has traditionally focused on pharmacologic therapies, particularly opioids, pain experts, clinical guidelines, and patients living with cancer increasingly support the use of non-pharmacologic therapies (including mind-body modalities such as distraction, mindfulness, and cognitive behavioral therapy) to mitigate pain and potentially reduce pain medication needs. Virtual reality (VR), a rapidly evolving technology that immerses the user in pleasant, virtual environments, has been shown to lower different forms of acute and chronic pain syndromes, but has not been developed specifically to improve chronic cancer pain. The long-term goal of the investigators is to develop and disseminate a patient-centered, patient-driven VR intervention that significantly improves the chronic cancer pain experience. Towards this end, they propose a multi-phase project involving active patient stakeholder input and an iterative design process that will achieve the following Specific Aims: Aim 1 - to identify patient perceptions around chronic cancer pain experiences and management strategies; Aim 2 - to develop a highly feasible, acceptable, usable, safe VR prototype enabling patient-directed management of cancer pain; Aim 3 - to conduct a trial to assess prototype feasibility, acceptability, usability, and safety. Completion of this project will lead towards development of a scalable VR intervention to mitigate pain that has potential to dramatically improve quality of life and clinical outcomes in patients living with chronic cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* living with active cancer diagnosis (any solid tumor type)
* report chronic cancer pain (≥3 months) with baseline severity moderate-severe (i.e., self-report pain score (SRPS) ≥4/10, where 0=no pain, 10=worst pain)
* prescribed chronic opioid therapies (may be long-acting formulations, short-acting formulations, or both)

Exclusion Criteria:

* history of intractable nausea/vomiting, motion sickness, seizures/epilepsy, and/or cranial structure abnormalities preventing VR headset use
* moderate-severe pain of non-cancer etiology (e.g., chronic lumbago)
* enrolled in another pain study
* unable to complete surveys in English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | From enrollment to end of treatment at 7 days
  >70% of participants completing the prescribed use of VR headset daily (≥10 minutes) for one week

SECONDARY OUTCOMES:
Acceptability | Collected at end of 7 days participation
  Technology Acceptance Model questionnaire
Usability | Collected at end of 7 day participation
  System Usability Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Groninger, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Georgetown Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided